CLINICAL TRIAL: NCT03626818
Title: The Impact of Neurocognitive Function in Patients With Multiple Brain Metastases Receiving Whole Brain Radiation Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1703
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-02

CONDITIONS: Brain Metastases
Keywords: WBRT; NCT
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NCF group: The patients have received 10 daily fractions of 3 Gy WBRT. Following WBRT treatment, subjects were assessed at each visit for NCT according to the Hopkins Verbal Learning Test-Revised(HVLT-R),Mini-Mental Status Examination(MMSE) and Quality Of Life measurements(QOL,Questionnaire-QLQC30).These tests was administered by trained and certified nurses or clinical research associates at baseline,6th week, 3rd, 6th, 9th, 12th month, and every 6 months until PS> 2 or intracranial tumor progression.

SUMMARY:
Brain metastases (BM), occurring in 10-30% of adult cancer patients, are an important cause of morbidity and mortality.The prognosis of patients with BM is generally poor, with a median survival time of 2-6 months. Whole-brain radiation therapy (WBRT) has been advocated as the primary treatment for metastatic brain cancer. WBRT injures small cerebral vasculature and neuropil,effects linked to imaging-defined white matter changes. However, information on the neurocognitive function(NCF) impact of WBRT in BM patients is also limited.This study aims to explore and evaluate the impact of NCF in patients with multiple brain metastases receiving WBRT.

DETAILED DESCRIPTION:
Brain metastases (BM), occurring in 10-30% of adult cancer patients, are an important cause of morbidity and mortality.The prognosis of patients with BM is generally poor, with a median survival time of 2-6 months. Whole-brain radiation therapy (WBRT) has been advocated as the primary treatment for metastatic brain cancer. WBRT injures small cerebral vasculature and neuropil,effects linked to imaging-defined white matter changes. However, information on the neurocognitive function(NCF) impact of WBRT in BM patients is also limited.This study aims to explore and evaluate the impact of NCF in patients with multiple brain metastases receiving WBRT.All patients were assessed at each visit for NCF according to the Hopkins Verbal Learning Test-Revised(HVLT-R),Mini-Mental Status Examination(MMSE) and Quality Of Life measurements(QOL,Questionnaire-QLQC30) .

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven solid tumor malignancy.
2. Brain MRI within 1 month of enrolment, at least three metastatic lesions in the brain (of which at least one had to be measurable according to Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1).
3. Males or females aged ≥18 years, < 75 years.
4. had an Eastern Cooperative Oncology Group (ECOG) performance-status score from 0 to 2.
5. A life expectancy of at least 3 months.
6. Adequate organ function according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0
7. Subjects did not receive other treatments such as cytotoxic drugs, radiotherapy (non-brain metastases) or surgery within 2 weeks.
8. Patients must have ability and general health that permits completion of the study requirements and required follow up.
9. Patients must be willing to complete NCF and QOL assessments at pre-specified time points outlined in the protocol.
10. Signed written informed consent

Exclusion Criteria:

1. Prior radiation therapy to the brain.
2. Radiologically or pathologically confirmed metastases in the spinal cord or meninges.
3. Taking sedatives and hypnotics, phenytoin, carbamazepine, rifampin, and barbiturate.
4. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, hepatic, renal, or metabolic disease).
5. Subjects suffered from dementia, mental illness and other serious cognitive dysfunction.

6.The patient's brain radiation dose needs to be increased. 7.Inability to comply with protocol or study procedures. 8.A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.

9.Pregnant female. 10.Breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple brain metastases will be referred through the department of Neurosurgery,Medical Oncology and Radiation-oncology at Guangdong General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Delayed recall deterioration rate(HVLT-R) | At 6 month

SECONDARY OUTCOMES:
Change in delayed recall(HVLT-R) | At 6th week, 3rd, 9th, 12th month
Change in recall(HVLT-R) | At 6th week, 3rd, 6th, 9th, 12th month
Change score(MMSE) | At 6th week, 3rd, 6th, 9th, 12th month
Change score(QLQBN20) | At 6th week, 3rd, 6th, 9th, 12th month
Intracranial progression-free survival for patients with different Graded Prognostic Assessment scores | At baseline,6th week, 3rd, 6th, 9th, 12th month, and every 6 months until Performance Status> 2 or intracranial tumor progression
Overall survival for patients with different GPA scores | At baseline,6th week, 3rd, 6th, 9th, 12th month, and every 6 months until PS> 2 or intracranial tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Yi Pan, Dr., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital & Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No